CLINICAL TRIAL: NCT03293875
Title: Adaptation and Implementation of Project Encuentro in the U.S.-Mexico Border
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City University of New York (Other)
Collaborators: Alliance of Border Collaboratives (Unknown); Programa Compañeros (Unknown)
Responsible Party: Principal Investigator, Julia Lechuga, Associate Professor, Hunter College of City University of New York
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 1U01MD010657-01 (NIH)
Record Dates: First submitted 2016-12-07; First posted 2017-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: HIV
Keywords: HIV Risk Reduction, Drug Use, Sexual Behavior, People who Inject Drugs, US-Mexico Border
MeSH Terms: conditions — Sexual Behavior

STUDY DESIGN:
Intervention Model Description: Quasi-experimental with sequential self-selective exposure to intervention
Masking Description: No Masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Social network HIV testing (Other): Participants will receive an HIV test
  Interventions: Behavioral: Social Network HIV Testing
- Peer network intervention (Other): Participants will receive psychoeducational sessions
  Interventions: Behavioral: Peer Network Intervention
- Community Events (Other): Participants will attend community events
  Interventions: Behavioral: Community Events

INTERVENTIONS:
Behavioral: Community Events — The coalitions in collaboration with CABs and peer leaders in their respective cities convened community meetings and events and invited PWID who had participated in other intervention components, who were receiving services at the partner organizations, and members at-large to participate. Events and meetings were advertised at the partner organizations offices, by staff during delivery of harm reductions supplies at places where PWID congregated to use drugs, and through social media. Events and meetings took place at community venues including parks, neighborhood gathering spaces, and at organizations. Events covered topics about HIV, sexual health, and human rights and included health fairs.
  Arms: Community Events
Behavioral: Social Network HIV Testing — The social network HIV testing intervention consisted of offering rapid HIV tests to PWID using a social network referral methodology.
  Arms: Social network HIV testing
Behavioral: Peer Network Intervention — Two peer leaders will be selected from each city to deliver the intervention sessions. Peer leaders will recruit drug users they know who will be asked, in turn, to recruit other drug users in their networks. Peer leaders will deliver the intervention to 300 drug users (150 per border city) in cycles composed of small social networks of 5-6 PWID.
  Arms: Peer network intervention

SUMMARY:
The proposed project is a research collaboration between the University of Texas at El Paso, The Alliance for Border Collaboratives in El Paso, Texas and Programa Companeros in Juarez City, Mexico to adapt, implement, and evaluate a multi-level community-based HIV prevention intervention (Project Encuentro). The intervention will target people who inject drugs (PWID) and consists of: 1) A social network HIV testing component, 2) a peer network psychoeducational intervention, and 3) community events. The intervention was developed in an area severely affected by violence and stigma towards people who use drugs (PWUD), El Salvador, which makes it particularly suitable for adaptation to meet the needs of PWUD living in the proposed intervention site, the U.S.-Mexico border. The proposed intervention site also has been severely affected by violence which has curtailed any prior attempts to reduce the risk of HIV acquisition among PWUD. Violence has worsened structural factors which affect HIV risk such as, increasing police persecution, stigma and reducing access to harm reduction resources. The investigators will engage in formative research to understand the context of HIV risk for PWID in the border region post violence and adapt the intervention accordingly. Findings will allow the investigators to tailor intervention components to meet the needs of PWID in the region. Subsequently, the investigators propose to test intervention effectiveness and evaluate implementation barriers and facilitators. To accomplish study aims a mixed qualitative, quantitative approach will be employed. The investigators will begin with a formative phase by conducting in-depth interviews with PWID (n = 40) living in the region to understand how the context of drug use and HIV risk changed as a result of the violence and will administer a social network survey (n = 200) to characterize the configuration of risk networks. Findings will yield the necessary information to culturally adapt the intervention to meet the needs of PWID in the region and will help the investigators focus recruitment efforts where the riskiest networks are located. After the intervention is adapted with the help of the community advisory boards and the community coalitions, the investigators will implement the intervention and will assess the effectiveness and reach via 3 waves of cross-sectional surveys administered to PWID (n=600). The investigators will assess the process of implementation by conducting ethnographic field notes of all intervention activities including community engagement and community advisory board and coalition meetings. The investigators will assess the fidelity and quality of the intervention. Lastly, the investigators will conduct key informant interviews with key stakeholders involved in the project and interviews and observations will be coded to reflect key systems factors related to successful implementation of intervention components in two intervention sites (El Paso, Texas and Ciudad Juarez, Mexico). Findings will be significant as the investigators will be conducting parallel research on the effectiveness of interventions for Latino PWUD in two very different contexts: El Salvador and the U.S-Mexico border. Findings will elucidate implementation challenges and barriers and such information can then be used to assess the effectiveness of diverse implementation strategies in organizations working to serve the needs of Latino PWUD.

DETAILED DESCRIPTION:
The intervention framework of the proposed Intervention informs the study approach and aim of exerting change at multiple levels, through community based approaches. At the individual level, the intervention components will target reductions in behaviors that increase HIV acquisition and at the structural level, reduce HIV stigma. At the individual level, the investigators propose to modify peer normative beliefs around engagement in behaviors that place individuals at risk of HIV including normative behavior around risky sexual encounters and injection drug use behaviors. Strategies to be employed in each intervention component are delineated below.

Social Network HIV Testing. To prepare for the rolling-out of the social network HIV testing component, the investigators will convene a two day training with partner organizations from both sides of the border to train staff on the social network referral methodology. Research staff will initiate the recruitment of seeds by recruiting four to six seeds per city. Counselors, at the partner organizations, will begin by administering a rapid HIV test and provide pre and post-test counseling to seeds. Counselors, who will be trained in the social network assessment methodology, will then ask seeds to list other PWID in their social network who they believe are at risk of contracting HIV. Counselors will then provide participants with 3 coupons to recruit identified network members for an HIV test. Referred participants who engage in high-risk behavior will be also provided with 3 coupons to refer their own network members for an HIV test. Whenever social network HIV testing rates slow, research staff will re-seed in the communities to begin the recruitment process again. Counselors will make appointments for all participants who test positive for confirmatory HIV testing at the respective local governmental health care institutions. A research staff will follow-up with HIV positive participants to engage them in care. Throughout the duration of the project, monthly meetings will be convened between research staff involved in the project to ascertain that procedures are being followed and retrain if the need arises. The social network component of the intervention will continue throughout the duration of the study. Fidelity will be monitored by the partner organizations who have extensive experience delivering HIV testing.

The Peer Network Intervention. Two peer leaders will be selected from each city to deliver the intervention sessions. Eligibility criteria will be being former PWID, having extensive contacts, high degree of trust among peers, and motivation and demonstrated ability to work fixed hours. Training sessions, in collaboration with partner organization, will be conducted to train peer leaders over the course of two weeks during ten training sessions lasting 3 hours per session. Peer leaders will be trained in the curriculum as well as in psychosocial theory as the basis for behavioral interventions, interactive group management, HIV risk reduction, effective instruction for role-plays, and social network recruitment methods. Peer leaders will recruit PWID they know who will be asked, in turn, to recruit other PWID in their networks. If this initial contact is unable to recruit network members, peer leaders will select other initial contact. Peer leaders will deliver the intervention to 300 PWID (150 per border city) in cycles composed of small social networks of 5-6 PWID. Four intervention cycles will be held per month and will consist of 3 consecutive sessions of 2 hours in duration delivered in the early afternoon. Peer leaders will be expected to comply with a fixed work schedule of 10 hours per week and will be asked to actively recruit social networks for each intervention cycle. The peer network intervention will have the following structure. The first session of the intervention will cover training in social contexts of risk and strategies to avoid them through role plays, techniques for harm reduction for injection drug use, and available community resources to deal with substance abuse. The second session will provide information about HIV and Sexually Transmitted Diseases through games, didactic sessions, and exercises to rank the risk of contracting HIV from various behaviors, negotiation skills for condom use in situations of high risk such as exchange of sex for drugs. The third session will consist of training in advocacy and sexual rights and establishment of a personal and social network risk reduction plan. Ethnographers will be trained to document the process of delivery such as number of participants per intervention cycle. Research staff will attend intervention sessions to assess intervention fidelity. Weekly meetings will be held with peer leaders and research staff to discuss problems, solutions.

Community-Wide Events. The community coalition in collaboration with the CAB and peer leaders will be asked to plan and convene meetings and implement events including health fairs at the community level with PWID to deliver health services and information on topics such as drug use prevention and treatment, HIV and risk reduction skills, and other issues affecting the HIV risk of communities such as persecution of PWID by police, human rights violations, and sexual violence. They will identify experts on topics identified and invite them as guest speakers. Fidelity will be assessed primarily assessed through process documentation (attendance logs, record-keeping) of event activities.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old
* able to give informed consent
* injected drugs in the last month
* engaged in sexual risk behavior in the last 3 months

Exclusion Criteria:

* under 18 years of age
* unable to give informed consent
* not able to provide informed consent
* did not inject drugs in the last month
* did not engage in sexual risk behavior in the last 3 months
* does not engage in sexual risk behavior

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 840 (Actual)
Dates: Start 2017-09-07 (Actual); Primary Completion 2022-08-24 (Actual); Study Completion 2022-12-10 (Actual)

PRIMARY OUTCOMES:
Condomless sex in exchange for drugs | 6 and 12 months post intervention delivery
  assessed by the ratio of number of sex acts in exchange for drugs and the number of those acts without a condom.

SECONDARY OUTCOMES:
Frequency of Drug Use | 6 and 12 moths post intervention delivery
  assessed by asking participants to report the number of days they used heroin and crack in the last 30 days.
Syringe Sharing | 6 and 12 moths post intervention delivery
  assessed by asking participants to report the frequency with which they injected with a syringe that had been used by another person and/or lent their used syringe to other people.

OTHER OUTCOMES:
Harm Reduction Behaviors | 6 and 12 moths post intervention delivery
  Mediator variable assessed by the number of harm reduction behaviors enacted in the last 30 days including condom use, use of sterile syringes, number of sexual partners, disseminating harm reduction information to peers, reducing substance use and injection with used syringes.
HIV stigma | 6 and 12 moths post intervention delivery
  Mediatior variable assessed by degree of agreement with statements conveying stigmatizing beliefs about HIV
Harm reduction norms | 6 and 12 moths post intervention delivery
  Process evaluation variable assessed with agreement with statements about perceived use of condoms, syringe sharing, and reduction in sexual partners by peers
Self-efficacy to enact harm reduction behaviors with peers | 6 and 12 moths post intervention delivery
  Process evaluation variable assessed with agreement with statements measuring degree of confidence in enacting harm reduction with peers including condom use and disinfecting syringes
Number of HIV tests | Monthly from date of intervention delivery through study completion
  A process and implementation evaluation measure assessed by the number of tests delivered during the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Julia Lechuga, PhD, Principal Investigator — City University of New York, School of Public Health; Rebeca Ramos, MPH, Study Director — Alliance of Border Collaboratives
Locations (2):
- Alliance of Border Collaboratives, El Paso, Texas, United States
- Programa Compañeros, Ciudad Juárez, Chihuahua, Mexico

IPD SHARING:
Plan to Share IPD: Yes
De-identified datasets and associated documentation (data dictionaries, annotated instruments, analytic code) will be deposited into a NIH-approved public repository within 12 months of the main publication
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: 9/14/2025
Access Criteria: De-identified datasets and associated documentation (data dictionaries, annotated instruments, analytic code) will be deposited into a NIH-approved public repository within 12 months of the main publication